CLINICAL TRIAL: NCT02826369
Title: Use of Compressed Sensing in Breast MRI
Acronym: COMPRIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-A00581-48
Record Dates: First submitted 2016-07-05; First posted 2016-07-11 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: Algorithms; Image Processing, Computer-Assisted/methods*; Magnetic Resonance Imaging/methods*; Data Compression; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3.0 Tesla in Magnetic Resonance Imaging (Experimental)
  Interventions: Other: 3.0 Tesla in Magnetic Resonance Imaging

INTERVENTIONS:
Other: 3.0 Tesla in Magnetic Resonance Imaging — Eligible patient will have a standard MRI. The images taken before 4min30 and after 6min after to the injection of gadolimium contrast medium will be carried out with the standard image acquisition.
  The images taken between 4min30 and 6min after the injection of gadolimium contrast medium will be carried out with the compressed sensing image acquisition.

SUMMARY:
Breast MRI is increasingly important in breast screening imaging. It is currently based on dynamic sequences after contrast injection whose temporal resolution must be less than 90 seconds with dynamic acquisitions at different times.

These curves profiles are designed to differentiate benign from malignant lesions. Recently, Mann et al, (2014) showed that increasing the temporal resolution of dynamic acquisitions; lesion enhancement curves over time were more accurate than the curves usually performed.

It seems necessary to work on sequences having better temporal resolution without compromising however spatial resolution.

ELIGIBILITY:
Inclusion Criteria:

* Patient to benefit a MRI in the assessment for a breast carcinoma
* Age >18 years old
* Assessment on 3.0 Tesla in Magnetic Resonance Imaging
* ECOG performance status ≤ 3
* Ability to provide an informed written consent form

Exclusion Criteria:

* Age < 18 years old
* Claustrophobia
* Contraindication to the injection of gadolinium contrast medium
* Contraindication to MRI
* Persons deprived of liberty or under supervision

Max Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2016-04-12 (Actual); Study Completion 2016-04-12 (Actual)

PRIMARY OUTCOMES:
Agreement between compressed sensing and standard image acquisition | 1 day
  Agreement between compressed sensing and standard image acquisition is defined by percentage of lesions detected by both modes of acquisitions

SECONDARY OUTCOMES:
Analysis of dammage contours | 1 day
  Analysis of lesions contours will be performed according to Bi-RADS classification
Image quality in compressed sensing acquisition | 1 day
  The image quality will be evaluated using a quality scale

CONTACTS AND LOCATIONS:
Overall Officials: OLDRINI Guillaume, MD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No